CLINICAL TRIAL: NCT03915821
Title: Memory Changes in Patients With Major Depression Disorder Treated With Electroconvulsive Therapy
Brief Title: Memory Changes in Patients With Major Depression Disorder Treated With ECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Nabiel Abd-Elhakeem Metawlly, Resident Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Memory Changes with ECT
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed as major depression according to DSM V (Experimental): All patients presented with major depression disorder not received ECT previously within 6 monthes, admitted to the study site ( Psychiatry department, in Assiut University Hospital, Assiut, Egypt). They Fulifilled will be recruited within 6 monthes duration .
  The patients classified into group A comprised that will be treated with Unipolar ECT, and group B comprised that will be treated Biploar ECT.
  Interventions: Device: ECT

INTERVENTIONS:
Device: ECT — Electroconvulsive therapy was administered by using bidirectional constant current, brief-pulse devices. During the procedure, the patients were sedated using propofol or thiopenthal. Succinylcholine (1 mg/kg) was used as muscle relaxant, and glycopyrrolate (0.2 mg) or atropine was used as an anticholinergic agent when necessary. The mean charges were 351 (SD, 143) mC for the unilateral electrode placement group, 417 (SD, 192) mC for the bitemporal electrode placement group and 260 (SD, 76) mC for the bifrontal electrode placement group, (Brus, Ole MSc, 2017).
  The average course of treatment for depression is 6 to 12 treatments, but some patients may require as many as 20 treatments,

SUMMARY:
The basic memory changes (impairment) present in patients with major depression and the influence of the treatment with ECT.

DETAILED DESCRIPTION:
Current literature provides insufficient information on the degree of cognitive impairment during and after electroconvulsive therapy (ECT), mostly due to the fact that applied tests lacked sensitivity and flexibility. Our goal was to evaluate cognitive functioning in adult depressed patients treated with bi & uni lateral & ECT, using tests sensitive for detection of possible acute and medium-term memory changes.(9) Major depressive disorder (MDD) is estimated to affect around 16 million Americans (Substance Abuse and Mental Health Services Administration [SAMHSA], 2013) and, according to the World Health Organization, is the leading cause of disability worldwide (World Health Organization 2012). Among In the U.S. workforce, the prevalence of MDD has been estimated at 7.6% .(2) Electroconvulsive therapy (ECT) is an effective treatment for severe depression but entails cognitive adverse effects, particularly the effects on memory. ECT may cause a temporary deficit in the cognitive processes of information encoding, consolidation, and retrieval. Transient memory disturbances are regarded as an inevitable adverse effect of therapeutic convulsions. Various strategies have been tried to decrease the cognitive adverse effects while retaining the antidepressant effect, including the use of unilateral instead of bilateral electrode placement, changes in waveform, and reducing the electrical stimulus intensity, (4).

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as having major depression according to DSM V.
2. Patients aged (18-50 years) of both sexes.

Exclusion Criteria:

1. History or current evidence of systemic medical illness, e.g.: hepatic, renal, cardiovascular, endocrinal, metabolic disorders or others.
2. History or current evidence of any Neurological disease.
3. Pregnant females.
4. Co-morbid psychiatric disorders other than depression.
5. Patients with mental subnormality.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the subjective memory changes present in a sample of patients with major depression disorder who admitted to psychiatry unit and evaluation of memory changes following ECT treatment . | Baseline
  Reach the least level of side effects in memory of Recent treatment with ECT in patient with major depression.
  measurement tool: _ History taking and full general & neurological examination to exclude any neurological disease.
  * Minim Mental State Examination, (MMSE) (Appendix I)
  * All Scales will be taken at date of admission, and at discharge up to 15 days and after three months of discharge .
    * All patients will be subjected to full psychiatric history and examination. The results of the above mentioned laboratory, investigations will be included in future analysis and interpretation of patients' abnormal psychiatric findings.
Evaluate the subjective memory changes present in a sample of patients with major depression disorder who admitted to psychiatry unit and evaluation of memory changes following ECT treatment | Baseline
  * Hamiliton rate Scale for depression,(HAM-D) (Appendix II),before and after treatment with ECT.
  * All Scales will be taken at date of admission,and at discharge up to 15 days and after three months of discharge .
Evaluate the subjective memory changes present in a sample of patients with major depression disorder who admitted to psychiatry unit and evaluation of memory changes following ECT treatment | Baseline
  Memory scale (MONTREAL COGNITIVE ASSESSMENT. MOCA), (Appendix III) All Scales will be taken at date of admission,and at discharge up to 15 days and after three months of discharge .

CONTACTS AND LOCATIONS:
Locations (1):
- Neuropsychiatry & Neurosurgery Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1-American Psychiatric Association, Review; 2018 (http://www.aetna.com/cpb/medical/data/400_499/0445.htm). 2-Birnbaum, H. G., et, al,. (2010). Employer burden of mild, moderate, and severe major depressive disorder: Mental health services utilization and costs, and work performance. J Clin Psychiatry.27: 78-89. 3-Brus, et al Subjective Memory Immediately Following Electroconvulsive Therapy. The Journal of ECT: June 2017 - 33 : 2 - 96-103. 4-Brus, et, al, (2017) Subjective Memory Immediately Following Electroconvulsive ; Therapy, The Journal of ECT: June 33 : 2 - 96-103 5-Greenberg, et al, (2015). The economic burden of adults with major depressive disorder in the United States (2005 and 2010). Journal of Clinical Psychiatry, 76: 155-162. 6-Kessler, R. C. (2012). The costs of depression. Psychiatric Clinic of North America, 35:1-14. 7-Philip S. Wang Gregory Simon Ronald C. Kessler First published: 24 March 2006, https://doi.org/10.1002/mpr.139. 8-UK ECT Review Group (2003). Efficacy and safety of electroconvulsive therapy in depressive disorders: a systematic review and meta-analysis. Lancet. 2003- 361:799-808. 9-N. P. Maric: et,al, psychological medicine Volume 46, Issue 4 March 2016 , pp. 797-806